CLINICAL TRIAL: NCT06943742
Title: Non-Helium Magnetoencephalography for Clinical Management of Pediatric Brain Tumors : An Observational Cohort Study
Brief Title: Non-Helium Magnetoencephalography in Pediatric Brain Tumors
Status: Recruiting | Type: Observational
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Collaborators: Beijing X-Magtech Technology Limited (Unknown)
Responsible Party: Sponsor
Other Study IDs: 449A01
Record Dates: First submitted 2025-03-03; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-03

CONDITIONS: Pediatric Brain Tumor
Keywords: Magnetoencephalography; Pediatric Brain Tumor
MeSH Terms: interventions — Magnetoencephalography; Tomography, X-Ray Computed; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Magnetoencephalography plus Computed Tomography/Magnetic Resonance Imaging — Use Magnetoencephalography and Computed Tomography/Magnetic Resonance Imaging in the preoperative assessment of pediatric brain tumors.

SUMMARY:
This observational study aims to evaluate the effectiveness of magnetoencephalography (MEG) in the preoperative assessment of pediatric brain tumors, particularly in determining the extent of resection, and compare it with computed tomography (CT) and magnetic resonance imaging (MRI).

The main questions this study aims to answer are:

What is the consistency between MEG and CT/MRI in localizing pediatric brain tumors? What is the clinical efficacy of MEG in determining the extent of resection of pediatric brain tumors preoperatively?

Participants will:

Undergo both MEG and CT/MRI examinations for preoperative assessment, and the extent of tumor resection will be determined by the comprehensive results of the above examinations.

Be followed up with MEG and CT/MRI at 1, 3, and 6 months after surgery, along with neurological and quality-of-life assessments.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 3-18 years old;
* Clinically diagnosed with brain tumor;
* Capable of cooperating with magnetoencephalography evaluation and recording.

Exclusion Criteria:

* Patients with serious comorbidities or neurological or psychiatric disorders that affect magnetoencephalography examination.
* Patients using drugs that affect central nervous system function;
* Patients who are not suitable for surgical procedures;
* Patients with progressive neurological disorders.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients of Guangzhou Women and Children's Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Consistency in Tumor Localization Between Magnetoencephalography (MEG) and Computed Tomography/Magnetic Resonance Imaging (CT/MRI) (Kappa Coefficient) | From enrollment to 12 months after surgery.
  The primary outcome will measure the agreement between MEG and CT/MRI (gold standard) in localizing pediatric brain tumors. Consistency will be quantified using the Kappa coefficient (κ), with sensitivity and specificity calculated for MEG against CT/MRI. Data will be aggregated by comparing preoperative MEG localization results (e.g., tumor location categorized by brain regions) with CT/MRI findings. Statistical analysis will include calculation of κ values (95% confidence interval), sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) using SPSS version 27.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Women and Children's medical center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No